CLINICAL TRIAL: NCT00404573
Title: A Double-Blind, Placebo-Controlled Evaluation of the Safety and Efficacy of RGH-188 in the Acute Exacerbation of Schizophrenia
Brief Title: Study Evaluating RGH-188 in the Treatment of Patients With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RGH-MD-03
Record Dates: First submitted 2006-11-27; First posted 2006-11-29 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2008-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — cariprazine

INTERVENTIONS:
Drug: RGH-188

SUMMARY:
This is a study designed to evalute the safety and efficacy of RGH-188 in the treatment of acute schizophrenia. This study will be 10 weeks in duration; 6 weeks double-blind treatment, and 4 weeks safety follow-up. All patients meeting the eligibility criteria will be randomized to one of the three treatment groups--one of two doses of RGH-188 or placebo

ELIGIBILITY:
Inclusion Criteria:

* Male and female inpatients, 18-65 years of age, meeting DSM-IV-TR criteria for schizophrenia and having a Total Positive and Negative Syndrome Scale (PANSS) Score >=80 and <=120. A score >=4 on item P1 (delusions) or P3 (hallucinatory behavior) and a score of >=4 on item P2 (conceptual disorganization) or P6 (suspiciousness/persecution) of the PNASS

Exclusion Criteria:

* Patients with documented disease of the central nervous system that can interfere with the trial assessments, including but not limited to stroke, tumor, Parkinson's, organic brain disease, seizure disorder (except for febrile convulsions during infancy), chronic infection, or neurosyphilis; or patients who have suffered a traumatic brain injury resulting in significant impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2006-11; Primary Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
PANSS Total Score

SECONDARY OUTCOMES:
CGI-S

CONTACTS AND LOCATIONS:
Locations (1):
- For information regarding investigative sites, contact Forest Professional Affairs, St Louis, Missouri, United States

REFERENCES:
- [Derived] Laszlovszky I, Barabassy A, Nemeth G. Cariprazine, A Broad-Spectrum Antipsychotic for the Treatment of Schizophrenia: Pharmacology, Efficacy, and Safety. Adv Ther. 2021 Jul;38(7):3652-3673. doi: 10.1007/s12325-021-01797-5. Epub 2021 Jun 6. PMID 34091867
- [Derived] Barabassy A, Sebe B, Acsai K, Laszlovszky I, Szatmari B, Earley WR, Nemeth G. Safety and Tolerability of Cariprazine in Patients with Schizophrenia: A Pooled Analysis of Eight Phase II/III Studies. Neuropsychiatr Dis Treat. 2021 Apr 7;17:957-970. doi: 10.2147/NDT.S301225. eCollection 2021. PMID 33854317
- [Derived] Earley W, Durgam S, Lu K, Laszlovszky I, Debelle M, Kane JM. Safety and tolerability of cariprazine in patients with acute exacerbation of schizophrenia: a pooled analysis of four phase II/III randomized, double-blind, placebo-controlled studies. Int Clin Psychopharmacol. 2017 Nov;32(6):319-328. doi: 10.1097/YIC.0000000000000187. PMID 28692485